CLINICAL TRIAL: NCT03701529
Title: Effect of Anesthetic Agents (Propofol, Sevoflurane) on Optic Nerve Sheath Diameter(ONSD) in Patients Undergoing Robot-assisted Laparoscopic Gynecology Surgery
Brief Title: Effect of Anesthetic Agents on Optic Nerve Sheath Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-09-004
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-01

CONDITIONS: Uterus Myoma; Uterine Cancer
MeSH Terms: conditions — Myofibroma; Uterine Neoplasms | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Experimental): 1.5-2.5 vol% of sevoflurane is used for maintenance of anesthesia.
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): 2-5 mcg/ml of propofol is used continuously for maintenance of anesthesia using target-controlled infusion system.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — 1.5-2.5 vol % sevoflurane is used for maintenance of anesthesia.
  Other Names: sevoflurane anesthesia
  Arms: Sevoflurane
Drug: Propofol — 2-5 mcg/ml of propofol is used for maintenance of anesthesia.
  Other Names: propofol anesthesia
  Arms: Propofol

SUMMARY:
The present study is to evaluate the effect of anesthetic agents ( propofol , sevoflurane) on intracranial pressure of female patients undergoing laparoscopic-robotic surgery.

DETAILED DESCRIPTION:
Anesthetic agents (propofol and sevoflurane)have different effect on intracranial pressure. Sevoflurane when used over 0.5 minimum alveolar concentration, dilates intracranial vasculature and increases intracranial pressure. On the other hand, propofol decreases intracranial blood pressure and intracranial pressure is maintained or decreases.

Optic nerve sheath diameter is a feasible diagnostic tool in evaluating intracranial pressure. Female patients undergoing robot-assisted laparoscopic hysterectomy or myomectomy are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* female patients undergoing robot-assisted laparoscopic hysterectomy or myomectomy

Exclusion Criteria:

* history of brain hemorrhage or brain infarction
* liver disease or end stage renal disease
* glaucoma or any signs of increased intraocular pressure
* combined wtih other types of operation
* patient refusal
* weight less than 40 kg or over 100 kg

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
difference of optic nerve sheath diameter | During the operation.
  optic nerve sheath diameter is measured using sonographic probe. (10 minutes after induction of anesthesia/ 5 minutes after pneumoperitoneum and trendelenburg position / 20 minutes after pneumoperitoneum and trendelenburg position / 40 minutes after pneumoperitoneum and trendelenburg position / skin closure)

CONTACTS AND LOCATIONS:
Overall Officials: Choi Eun-Mi, Professor, Study Chair — Kangnam Sungshim Hospital
Locations (1):
- Kangnam Sungshim Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No